CLINICAL TRIAL: NCT06373627
Title: Procedural Pain Management by Multimodal Sedation Analgesia Combining Hypnosis in Children With Congenital Heart Disease: a Randomized Non-inferiority Trial.
Brief Title: Procedural Pain Management by Multimodal Sedation Analgesia Combining Hypnosis in Children With Congenital Heart Disease
Acronym: PEACE-HYPNO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-A00534-43
Record Dates: First submitted 2024-04-10; First posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Procedural Pain; Congenital Heart Disease; Heart Surgery; Hypnosis
Keywords: Congenital Heart Disease; Procedural Pain; Intrathoracic drain; Hypnosis; Pain controlled; Heart surgery
MeSH Terms: conditions — Pain, Procedural; Heart Defects, Congenital | interventions — Hypnosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypnosis (Experimental): Hypnosis + MEOPA + direct intravenous Ketamine (0.3 mg/kg) In the event of insufficient analgesia or failure of hypnosis, a 2nd dose of ketamine (0.3 mg/kg) may be administered.
  Interventions: Other: Hypnosis; Drug: Medications used in addition to hypnosis
- Conventional sedation-analgesia (Active Comparator): MEOPA + direct intravenous Ketamine (0.5 mg/kg) + direct intravenous Midazolam (50 µg/kg) In accordance with current service protocol.
  Interventions: Drug: Conventional medications used for sedation-analgesia

INTERVENTIONS:
Other: Hypnosis — A hypnosis session takes place in 3 stages:
  * An induction stage, where we move from an ordinary state of consciousness to a modified state of consciousness through dissociation.
  * A work phase to deepen the hypnotic trance. This phase is fueled by the construction of suggestions and metaphors, analogous to those of the patient in pain.
  * Finally, a return to the ordinary state of consciousness through re-association with the patient.
  Arms: Hypnosis
Drug: Conventional medications used for sedation-analgesia — MEOPA + intravenous ketamine (0.5 mg/kg) + intraveinous midazolam (50µg/kg)
  Arms: Conventional sedation-analgesia
Drug: Medications used in addition to hypnosis — MEOPA + intravenous ketamine (0.3 mg/kg)
  Arms: Hypnosis

SUMMARY:
The aim of this prospective randomized controlled trial is to evaluate therapeutic hypnosis as a co-analgesia in thoracic drain removal in children with congenital heart disease. The hypothesis of this study is that therapeutic hypnosis combined with a minimal effective dose of medicated and inhaled sedation-analgesia is not inferior to higher doses of sedation-analgesia usually employed. This would make possible the reduction of cumulative dose of sedative medication and their side effects.

DETAILED DESCRIPTION:
Pain and anxiety are common in children with congenital heart disease. They are at risk to develop impaired pain signal processing, and tolerance to opioids and benzodiazepines due to repeated exposure.

Removal of thoracic drains is a standard procedure following cardiac surgery in patients with congenital heart disease. This procedure is usually performed after multimodal sedation-analgesia (intraveinous and inhalation drugs). However, the drugs used (ketamine and midazolam) can have significant side-effects, such as respiratory and circulatory depression.

A few studies have shown the efficacy of therapeutic hypnosis and distractive methods in children, but with a low level of evidence, unlike in adults.

However, none of these studies has evaluated therapeutic hypnosis in children with congenital heart disease.

Hypnosis would be an additional way of better controlling procedural pain, without the side effects of medication. This would reduce the dose of analgesic drugs and improve the pain experience.

The aim of PEACE-Hypno is to evaluate therapeutic hypnosis as a co-analgesic way of thoracic drain removal in children with congenital heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ⩾ 6 years and <18 years.
* Postoperative cardiac surgery patients with intrathoracic drains (pleural or mediastinal).
* Patients affiliated with or benefiting from a social security or similar scheme.
* Oral consent obtained from minor children
* Written consent from the minor's legal representatives

Exclusion Criteria:

* Psychomotor retardation, cognitive/psychiatric impairment preventing self-assessment of pain
* Absence of at least 1 legal representative of the minor child
* French not understood

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 104 (Estimated)
Dates: Start 2024-05-02 (Estimated); Primary Completion 2025-05-02 (Estimated); Study Completion 2025-05-03 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome : Pain evaluation by VAS self-assessment | VAS will be measured 5 minutes before the start of the procedure (T0) and at the end of the procedure (T1) to assess the average pain intensity during drain removal.
  The use of therapeutic hypnosis in addition to a minimal effective dose of intravenous and inhaled sedation-analgesia does not change level of pain generated by conventional sedation-analgesia during intrathoracic drain removal in children aged 6 to 18 years with congenital heart disease, self-assessed by VAS.

SECONDARY OUTCOMES:
Hetero-assessment by FLACC scale of the pain during the intrathoracic drain removal | Scoring of the FLACC scale by the evaluator through study completion (up to1 year), blinded to the allocation arm, based on the video recorded during the procedure.
  The use of therapeutic hypnosis in addition to a minimal effective dose of intravenous and inhaled sedation-analgesia generates non-inferior pain to that generated by conventional sedation-analgesia during intrathoracic drain removal in children aged 6-18 years with congenital heart disease, in hetero-assessment by FLACC by a blinded assigning arm assessor.
Maximum heart rate | The maximum heart rate is measured during the intrathoracic drain removal, through the beginning to the end of procedure
  Comparison between the two groups of the maximum heart rate during intrathoracic drain removal, measured continuously on a monitor.
Cumulative doses of intravenous analgesics | Cumulative doses of intravenous analgesics refer to drugs administered from the beginning to the end of the procedure.
  Comparison between the two groups of the cumulative doses of Ketamine and Midazolam used during the procedure.
Respiratory depression | The number of respiratory depression is measured during the intrathoracic drain removal, through the beginning to the end of procedure.
  Comparison between the two groups of the number of episodes of respiratory depression corresponding to a respiratory rate of less than 10/min, measured continuously using the scope.
Parental satisfaction using Visual Analogic Scale (VAS) | Parents evaluate their satisfaction the day after the procedure (D+1), with a minimal value of 0/10 (e.g no satisfaction), and a maximal value of 10/10 (maximal satisfaction)
  Parents evaluate their satisfaction about the procedure, using a VAS self-assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Edouard CHAMBON, Principal Investigator — Fondation Hôpital Saint-Joseph

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Staveski SL, Boulanger K, Erman L, Lin L, Almgren C, Journel C, Roth SJ, Golianu B. The Impact of Massage and Reading on Children's Pain and Anxiety After Cardiovascular Surgery: A Pilot Study. Pediatr Crit Care Med. 2018 Aug;19(8):725-732. doi: 10.1097/PCC.0000000000001615. PMID 29912070
- [Background] Krauss B, Green SM. Procedural sedation and analgesia in children. Lancet. 2006 Mar 4;367(9512):766-80. doi: 10.1016/S0140-6736(06)68230-5. PMID 16517277
- [Background] Birnie KA, Noel M, Chambers CT, Uman LS, Parker JA. Psychological interventions for needle-related procedural pain and distress in children and adolescents. Cochrane Database Syst Rev. 2018 Oct 4;10(10):CD005179. doi: 10.1002/14651858.CD005179.pub4. PMID 30284240
- [Background] Accardi MC, Milling LS. The effectiveness of hypnosis for reducing procedure-related pain in children and adolescents: a comprehensive methodological review. J Behav Med. 2009 Aug;32(4):328-39. doi: 10.1007/s10865-009-9207-6. Epub 2009 Mar 3. PMID 19255840
- [Background] Geagea D, Tyack Z, Kimble R, Polito V, Ayoub B, Terhune DB, Griffin B. Clinical Hypnosis for Procedural Pain and Distress in Children: A Scoping Review. Pain Med. 2023 Jun 1;24(6):661-702. doi: 10.1093/pm/pnac186. PMID 36448690
- [Background] Chester SJ, Stockton K, De Young A, Kipping B, Tyack Z, Griffin B, Chester RL, Kimble RM. Effectiveness of medical hypnosis for pain reduction and faster wound healing in pediatric acute burn injury: study protocol for a randomized controlled trial. Trials. 2016 Apr 29;17(1):223. doi: 10.1186/s13063-016-1346-9. PMID 27129580
- [Background] Stinson JN, Kavanagh T, Yamada J, Gill N, Stevens B. Systematic review of the psychometric properties, interpretability and feasibility of self-report pain intensity measures for use in clinical trials in children and adolescents. Pain. 2006 Nov;125(1-2):143-57. doi: 10.1016/j.pain.2006.05.006. Epub 2006 Jun 13. PMID 16777328
- [Background] Rodrigues VBM, Costa LR, Correa de Faria P. Parents' satisfaction with paediatric dental treatment under sedation: A cross-sectional study. Int J Paediatr Dent. 2021 May;31(3):337-343. doi: 10.1111/ipd.12661. Epub 2020 Jun 21. PMID 32412090
- [Background] Crellin DJ, Harrison D, Santamaria N, Babl FE. Systematic review of the Face, Legs, Activity, Cry and Consolability scale for assessing pain in infants and children: is it reliable, valid, and feasible for use? Pain. 2015 Nov;156(11):2132-2151. doi: 10.1097/j.pain.0000000000000305. PMID 26207651
- [Background] Crellin D, Harrison D, Santamaria N, Babl FE. Comparison of the Psychometric Properties of the FLACC Scale, the MBPS and the Observer Applied Visual Analogue Scale Used to Assess Procedural Pain. J Pain Res. 2021 Mar 31;14:881-892. doi: 10.2147/JPR.S267839. eCollection 2021. PMID 33833566
- [Background] Abdolkarimi B, Zareifar S, Golestani Eraghi M, Saleh F. Comparison Effect of Intravenous Ketamine with Pethidine for Analgesia and Sedation during Bone Marrow Procedures in Oncologic Children: A Randomized, Double-Blinded, Crossover Trial. Int J Hematol Oncol Stem Cell Res. 2016 Oct 1;10(4):206-211. PMID 27928474
- [Background] Chiaretti A, Ruggiero A, Barbi E, Pierri F, Maurizi P, Fantacci C, Bersani G, Riccardi R. Comparison of propofol versus propofol-ketamine combination in pediatric oncologic procedures performed by non-anesthesiologists. Pediatr Blood Cancer. 2011 Dec 15;57(7):1163-7. doi: 10.1002/pbc.23170. Epub 2011 May 16. PMID 21584935
- [Background] Rayala S, Kyander M, Haridass V, Palat G, Strom A, Wiebe T, Brun E, Segerlantz M. Low-dose Oral Ketamine as a Procedural Analgesia in Pediatric Cancer Patients Undergoing Bone Marrow Aspirations at a Resource-limited Cancer Hospital in India. Indian J Palliat Care. 2019 Oct-Dec;25(4):501-507. doi: 10.4103/IJPC.IJPC_110_19. PMID 31673202
- [Background] Myles PS, Myles DB, Galagher W, Boyd D, Chew C, MacDonald N, Dennis A. Measuring acute postoperative pain using the visual analog scale: the minimal clinically important difference and patient acceptable symptom state. Br J Anaesth. 2017 Mar 1;118(3):424-429. doi: 10.1093/bja/aew466. PMID 28186223
- [Background] Luo D, Wan X, Liu J, Tong T. Optimally estimating the sample mean from the sample size, median, mid-range, and/or mid-quartile range. Stat Methods Med Res. 2018 Jun;27(6):1785-1805. doi: 10.1177/0962280216669183. Epub 2016 Sep 27. PMID 27683581
- [Background] Piaggio G, Elbourne DR, Pocock SJ, Evans SJ, Altman DG; CONSORT Group. Reporting of noninferiority and equivalence randomized trials: extension of the CONSORT 2010 statement. JAMA. 2012 Dec 26;308(24):2594-604. doi: 10.1001/jama.2012.87802. PMID 23268518
- [Background] Chanques G, Jaber S, Barbotte E, Verdier R, Henriette K, Lefrant JY, Eledjam JJ. [Validation of the french translated Richmond vigilance-agitation scale]. Ann Fr Anesth Reanim. 2006 Jul;25(7):696-701. doi: 10.1016/j.annfar.2006.02.017. Epub 2006 May 15. French. PMID 16698231
- [Background] Ely EW, Inouye SK, Bernard GR, Gordon S, Francis J, May L, Truman B, Speroff T, Gautam S, Margolin R, Hart RP, Dittus R. Delirium in mechanically ventilated patients: validity and reliability of the confusion assessment method for the intensive care unit (CAM-ICU). JAMA. 2001 Dec 5;286(21):2703-10. doi: 10.1001/jama.286.21.2703. PMID 11730446
- [Background] Sessler CN, Gosnell MS, Grap MJ, Brophy GM, O'Neal PV, Keane KA, Tesoro EP, Elswick RK. The Richmond Agitation-Sedation Scale: validity and reliability in adult intensive care unit patients. Am J Respir Crit Care Med. 2002 Nov 15;166(10):1338-44. doi: 10.1164/rccm.2107138. PMID 12421743